CLINICAL TRIAL: NCT03249870
Title: A Phase 2 Study of Inotuzumab Ozogamicin (INO) Combined to Chemotherapy in Older Patients With Philadelphia Chromosome-negative CD22+ B-cell Precursor Acute Lymphoblastic Leukemia
Brief Title: Study of Inotuzumab Ozogamicin Combined to Chemotherapy in Older Patients With Philadelphia Chromosome-negative CD22+ B-cell Precursor ALL
Acronym: EWALL-INO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Patrice Chevallier, MD, PhD, Nantes University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P16/11- EWALL INO; 2016-004942-27 (EudraCT Number)
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Acute Lymphoblastic Leukemia (ALL) - Philadelphia Chromosome (Ph)-Negative CD22+ B-cell Precursor (BCP)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia Chromosome | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inotuzumab ozogamicin (INO) (Experimental)
  Interventions: Drug: Inotuzumab ozogamicin (INO)

INTERVENTIONS:
Drug: Inotuzumab ozogamicin (INO) — INO schedule of administration is as follows:
  * First induction course: 0.8 mg/m² on day 1, 0.5 mg/m² on day 8, and 0.5 mg/m² on day 15
  * Second induction course: 0.5 mg/m² on day 1, and 0.5 mg/m² on day 8

SUMMARY:
The aim of the present EWALL-INO study is to confirm very promising results obtained with a combination of INO and mild chemotherapy in older de novo CD22+ B-ALL patients. For that purpose, safety and efficacy of a weekly INO administration combined to mild-intensity chemotherapy will be evaluated in a cohort of patients aged more than 55 years with newly diagnosed previously untreated Ph-negative (CD22+) BCP-ALL. Conversely to the MDACC miniHCVD-INO study and in order to lower the overall toxicity of the combination, INO will be given as part of the remission induction treatment phase during the first 2 treatment cycles only, in combination with corticosteroid, vincristine, cyclophosphamide and intrathecal prophylaxis only; then, all responding patients will received standard INO-free chemotherapy as consolidation and maintenance.

DETAILED DESCRIPTION:
INO schedule of administration will be as described in the refractory/relapsed INO-VATE study for the first cycle, with sequential day 1/8/15 doses of 0.8, 0.5 and 0.5 mg/m2, respectively. Reduced dose of INO will be used for the second and last cycle (0.5 mg/m2 on day 1/8). This was retained in order:

1. to minimize potential toxicities, including liver disorders and prolonged thrombocytopenia; and
2. to allow delivery of subsequent chemotherapy consolidations cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 55 years old,
* With confirmed diagnosis of BCP-ALL according to World Health Organisation (WHO) criteria expressing the CD22 antigen by flow cytometry (20% or more positive blast cells),
* Without central nervous system (CNS) involvement,
* Without BCR-ABL fusion by standard cytogenetics, Fluorescence In Situ Hybridization (FISH) analysis and/or RT-PCR,
* Previously untreated,
* Eligible to intensive chemotherapy, due to general health status,
* ECOG performance status ≤ 2,
* Patients must have the following laboratory values unless considered due to leukemia: AST and ALT ≤ 2.5 x upper the limit of normal (ULN); estimated GFR ≥ 50 mL/min using the MDRD equation; total and direct serum bilirubin ≤ 1.5 x ULN; electrolyte panel within normal ranges for the institution unless attributed to the underlying disease.
* Written informed consent obtained prior to any screening procedures.
* Eligible for National Health Insurance in France.

Exclusion Criteria:

* Concurrent therapy with any other investigational agent or cytotoxic drug,
* Prior documented chronic liver disease,
* Active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) or positive HIV serology,
* Female patients who are pregnant or breast feeding or patients of childbearing potential not willing to use a double barrier method of contraception during the study and for 3 months following the last dose of maintenance.
* Male patients whose sexual partner(s) are women of childbearing potential who are not willing to use a double barrier method of contraception, one of which includes a condom, during the study and for 3 months following the last dose of maintenance.
* Any of concurrent severe and/or uncontrolled medical condition, which could compromise participation in the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-12-28 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of overall survival (OS) | one year
  The primary objective of the trial is to assess overall survival (OS) observed at 1 year after administration of INO and chemotherapy in older Ph-negative BCP-ALL patients.

SECONDARY OUTCOMES:
Assessment of adverse events (AEs) | 3 months
  Type, duration and frequency of AEs up to 3 months of induction course 1 or 2
Rate of complete remission (CR / CRp) | 35 days
  CR/CRp response rate after INO-based induction course 1 and 2
Assessment of Minimal residual disease (MRD) | 35 days
  Flow cytometry and Ig-TCR MRD levels, after INO-based induction course 1 and 2 and impact on outcomes
Rate of early death | 100 days
  Early death (ED) rate at 30, 60 and 100 day from treatment initiation
Composite measure for Duration of response (DOR), Disease-free survival (DFS) and cumulative incidence of relapse (CIR) | one year
  Duration of response (DOR), Disease-free survival (DFS) and cumulative incidence of relapse (CIR)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice CHEVALLIER, MD, Principal Investigator — Nantes University Hospital
Locations (41):
- France (41):
  - CH Amiens sud, Amiens
  - CHU Angers, Angers
  - CH Victor Dupouy, Argenteuil
  - CH cote basque, Bayonne
  - CHU Besançon, Besançon
  - Hopital Avicenne, Bobigny
  - Hopital Duchenne, Boulogne-sur-Mer
  - CHU Caen, Caen
  - CH Rene Dubois, Cergy-Pontoise
  - CH metropole Savoie_ chambery, Chambéry
  - HIA Percy, Clamart
  - CHU Clermond Ferrand, Clermont-Ferrand
  - Hopital Mondor, Créteil
  - Hopital Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHU la Reunion, La Réunion
  - CH Versailles, Le Chesnay
  - CHU Limoges, Limoges
  - Centre Leon Berard, Lyon
  - IPC, Marseille
  - CH Meaux, Meaux
  - CH Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Centre Lacassagne, Nice
  - CHU Nice, Nice
  - CHU Nimes, Nîmes
  - CHR Orléans, Orléans
  - Hopital Necker, Paris
  - Hopital St Antoine, Paris
  - Hopital St Louis, Paris
  - CHU Haut Leveque, Pessac
  - CH Lyon Sud, Pierre-Bénite
  - CH Reims, Reims
  - CHU Pontchaillou, Rennes
  - CH Roubaix, Roubaix
  - Centre H Becquerel Rouen, Rouen
  - Institut de cancerologie, Saint-Priest-en-Jarez
  - CHU Strasbourg, Strasbourg
  - IUCT Oncopole, Toulouse
  - CH Valenciennes, Valenciennes
  - CHRU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chevallier P, Leguay T, Delord M, Salek C, Kim R, Huguet F, Hicheri Y, Wartiovaara-Kautto U, Raffoux E, Cluzeau T, Balsat M, Roth-Guepin G, Tavernier E, Lepretre S, Bilger K, Bergugnat H, Berceanu A, Alexis M, Doubek M, Brissot E, Hunault-Berger M, Lebon D, Turlure P, Chantepie S, Belhabri A, Wickenhauser S, Bastie JN, Cacheux V, Himberlin C, Banos A, Gardin C, Bonnet S, Plantier I, Pica GM, Escoffre-Barbe M, Boissel N, Dombret H, Clappier E, Rousselot P; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL) and the European Working Group for Adult Acute Lymphoblastic Leukemia (EWALL); European Working Group for Adult Acute Lymphoblastic Leukemia (EWALL). Inotuzumab Ozogamicin and Low-Intensity Chemotherapy in Older Patients With Newly Diagnosed CD22+ Philadelphia Chromosome-Negative B-Cell Precursor Acute Lymphoblastic Leukemia. J Clin Oncol. 2024 Dec 20;42(36):4327-4341. doi: 10.1200/JCO.24.00490. Epub 2024 Oct 17. PMID 39418626